CLINICAL TRIAL: NCT06175182
Title: A Comparison of Exercise Capacity, Arterial Stiffness, and Cognitive Function Between Adults With Cystic Fibrosis and Healthy Individuals
Brief Title: Assessment of Cognitive Function and Exercise Capacity in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Deniz Inal-Ince, Professor, Hacettepe University
Other Study IDs: GO 22/917
Record Dates: First submitted 2023-11-30; First posted 2023-12-18 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; exercise test; cognitive impairment; arterial stiffness
MeSH Terms: conditions — Cystic Fibrosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cystic fibrosis: No intervention
- healthy volunteers: No intervention

SUMMARY:
No studies in the literature have investigated the simultaneous effects of cognitive function, exercise capacity and arterial stiffness in adult patients with CF. The study aims to compare the cognitive function, exercise capacity, exercise muscle oxygenation, and arterial stiffness of adult patients with CF and healthy subjects.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) affects other body systems as well as the respiratory system. Patients with CF seem to have reduced exercise capacity, which is a major contributor to mortality rates. Changes in lung function, ventilatory dysfunction, and respiratory muscle function potentially contribute to exercise intolerance in CF. Both children and adults with CF exhibit neurocognitive dysfunction. Arterial stiffness is a predictor of cardiovascular events, including myocardial infarction, heart failure, and mortality. Individuals with CF exhibit an increase in arterial stiffness. However, no studies in the literature have investigated cognitive function, exercise capacity, and arterial stiffness coexistence in adult CF patients. The study aims to compare the cognitive function, exercise capacity, exercise muscle oxygenation and arterial stiffness in adult patients with CF and healthy subjects. Additionally, it will determine the relationship between cognitive function and arterial stiffness with exercise capacity and muscle oxygenation during exercise in adult patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with cystic fibrosis
* Being 18 years old and older
* Clinically stable condition
* Able to cooperate with the tests performed
* Volunteered to participate in the study

For the control group:

* Being 18 years old and older
* Volunteered to participate in the study

Exclusion Criteria:

* History of hospitalization or exacerbation in the last month.
* Chronic respiratory failure and long-term use of oxygen therapy
* Using noninvasive mechanical ventilator therapy
* Indication for lung transplantation
* Who had a lung transplant
* Forced expiratory volume in the first second (FEV1) value 30% and below
* CF-related diabetes
* Chronic liver disease
* Allergic bronchopulmonary aspergillosis
* Systemic steroid use
* History of diagnosed orthopedic or musculoskeletal problems affecting mobility
* Cardiovascular instability
* Serious psychiatric illness

For the control group:

* Known chronic or systemic disease
* Who did not volunteer to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 24 patients with cystic fibrosis will be included in patients group and 24 healthy individuals will be included in control group.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 6 minutes
  Exercise capacity is assessed using the 6-minute walk test (6MWT). The 6MWT is performed according to the criteria of the American Thoracic Society.
Arterial Stiffness Assessment | 20 minutes
  Arterial stiffness is determined using a oscillometric cuff device (Tel-O-Graph BT, I.E.M., Stolberg, Germany). Pulse wave velocity (PWV) and augmentation index (AIx) are measured by brachial pulse waves.
Cognitive Assessment- MoCA | 10 minutes
  Cognitive function is measured using the Montreal Cognitive Assessment (MoCA) test. The MoCA test is a questionnaire developed to evaluate different cognitive functions and mild cognitive impairment. The maximum score that an individual can obtain from the test is 30, and a score of 26 above is considered as mild cognitive impairment.
Cognitive Assessment-Mini Mental Test | 10 minutes
  Cognitive function is measured using the Mini Mental Test. A higher score indicates better cognitive function. The maximum score that an individual can obtain from the test is 30, and a score of 23 and above is considered as cognitive impairment.
Muscle Oxygenation Assessment | 10 minutes
  Muscle oxygenation (SmO2) is assessed using a measuring and monitoring device (Moxy Fortiori Desing LLC, Minnesota, USA).

SECONDARY OUTCOMES:
Body Composition | 5 minutes
  Body fat is measured using skinfold thickness assessment.
Pulmonary Function Test (forced vital capacity (FVC)) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses forced vital capacity (FVC).
Pulmonary Function Test (forced expiratory volume in the first second (FEV1)) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses forced expiratory volume in the first second (FEV1).
Pulmonary Function Test (FEV1/FVC) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses FEV1/FVC.
Pulmonary Function Test (peak flow rate (PEF)) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses peak flow rate (PEF).
Pulmonary Function Test (forced expiratory flow from 25-75% (FEF25-75%)) | 10 minutes
  Testing procedures is in accordance with the guidelines published by ATS/ERS. A portable spirometer is used for assessment. Pulmonary function testing assesses forced expiratory flow from 25-75% (FEF25-75%).
Respiratory Muscle Strength | 10 minutes
  Maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) are measured using a mouth pressure measuring device with personal antibacterial and antiviral disposable filters.
Peripheral Muscle Strength | 5 minutes
  Knee extensor muscle strength is measured utilizing a portable device.
Anxiety and Depression | 5 minutes
  The Hospital Anxiety and Depression scale (HADS) is used to evaluate anxiety and depression. Higher scores correspond to more anxiety and depression symptoms.
Physical Activity Assessment | 5 minutes
  Physical activity levels is assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-SF). The IPAQ requires respondents to estimate time spent in various levels of physical activity during the previous week. Scores for walking and moderate and vigorous activities are calculated as durations and frequencies multiplied by known metabolic equivalents per activity. The results for all activity-based items are summed for the total physical activity score. The participants were then categorized as inactive, minimally active and sufficiently active according to the IPAQ categorical classification.
Sleep Quality | 5 minutes
  Sleep quality is evaluated using the Pittsburgh Sleep Quality Index (PSQI). The scale total score is between 0 and 21. A total score of 5 and above indicates poor sleep quality.
Disease Specific Quality of Life | 8 minutes
  Disease-specific quality of life is evaluated using the Cystic Fibrosis Questionnaire-Revised (CFQ-R). The CFQ-R includes 50 items across 12 domains. Each domain is standardized on a 0-100 scale; higher scores indicate better quality of life.
General Health-Related Quality of Life | 5 minutes
  Health-related quality of life is assessed using the Nottingham Health Profile (NHP). It is a general QOL questionnaire designed to measure perceived health problems and the extent to which these problems affect normal daily activities. It consists of 38 items in six dimensions (energy level, pain, physical mobility, emotional reactions, social isolation, and sleep). The total score for each section is 0-100. High scores indicate worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)